CLINICAL TRIAL: NCT00237237
Title: Vildagliptin Compared to Pioglitazone in Combination With Metformin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2354
Record Dates: First submitted 2005-10-09; First posted 2005-10-12 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
Many people with type 2 diabetes cannot maintain target blood glucose levels when taking a single oral drug. The purpose of this study is to assess the long-term safety and effectiveness of vildagliptin, an unapproved drug, compared to that of pioglitazone in lowering overall blood glucose levels when added to metformin in people with type 2 diabetes not at target blood glucose levels on metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* On a stable dose of metformin as defined by the protocol
* Blood glucose criteria must be met
* Body mass index (BMI) in the range 22-45

Exclusion Criteria:

* History of type 1 diabetes
* Pregnancy or lactation
* Evidence of significant diabetic complications
* Serious cardiovascular events within the past 6 months
* Laboratory value abnormalities as defined by the protocol
* Known sensitivity to pioglitazone
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 77 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 588
Dates: Start 2005-10; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 52 weeks

SECONDARY OUTCOMES:
Adverse event profile after 52 weeks of treatment
Change from baseline in fasting plasma glucose at 52 weeks
Change from baseline in body weight at 52 weeks
Patients with endpoint HbA1c < 7% after 52 weeks
Patients with reduction in HbA1c >/= to 7% after 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Investigative Centers, Nuremberg, Germany

REFERENCES:
- [Result] Bolli G, Dotta F, Rochotte E, Cohen SE. Efficacy and tolerability of vildagliptin vs. pioglitazone when added to metformin: a 24-week, randomized, double-blind study. Diabetes Obes Metab. 2008 Jan;10(1):82-90. doi: 10.1111/j.1463-1326.2007.00820.x. Epub 2007 Nov 22. PMID 18034842